CLINICAL TRIAL: NCT02525887
Title: A Clinical Trial to Identify Genetic Variations That Affect The Ability of Patients To Metabolize Drugs Through Metabolic Pathways 2C19, 2C9, 2D6, 3A4, 3A5, Factor II, Factor V, MTHFR and VKORC1
Brief Title: Identify Genetic Variations That Affect The Ability of Patients To Metabolize Drugs Through Metabolic Pathways
Status: Terminated | Type: Observational
Why Stopped: Study cancelled
Sponsor: Bracane Company (Industry)
Collaborators: IFG Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: IFG201502-PGX
Record Dates: First submitted 2015-08-11; First posted 2015-08-18 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Disease; Endocrine System Disease; Cardiovascular Disease; Respiratory Tract Disease; CNS Metabolic Disorders
MeSH Terms: conditions — Chronic Disease; Endocrine System Diseases; Cardiovascular Diseases; Respiratory Tract Diseases; Brain Diseases, Metabolic | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observation — Observation and evaluation of care provided to patients that received DNA tests to determine metabolic pathways.

SUMMARY:
This observation will look at patient care decisions of the primary healthcare provider utilizing the results of the DNA testing of patients' metabolic pathways using 2C19, 2C9, 2D6, 3A4, Factor II, Factor V and MTHFR and VKORC1. Findings of the data collection will be published to optimize the benefits of pharmacogenomics testing and publish health outcomes.

DETAILED DESCRIPTION:
This study will analyze de-identified data from patients identified by the primary healthcare provider where a DNA sample has been collected; the medical history and medications at the time the DNA sample was collected; the date of the DNA pathway testing and the results. The study will collect and assess the patient data where the healthcare provider has explained the results of the DNA testing to the patient and made applicable changes in the healthcare plan based on the DNA pathway results. Patients will have returned to the healthcare provider after a minimum of ninety (90) days for follow-up to assess the outcome of the care plan changes started after the DNA results provided. This study will collect the healthcare provider will provide the outcomes of the healthcare plan changes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients age 18 or older
2. Prescribed at least one medication with in any of the metabolic pathways being assessed will be enrolled in the study.
3. Completed DNA testing for the pathways under review for this observation.

Exclusion Criteria:

1. Anticipated life expectancy less than 1 month.
2. Employee of the investigator, with direct involvement in the proposed study or other studies under the direction of the investigator, as well as immediate family members or the employee or primary care provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data from a total of approximately 10,000 adult male or female patients age 18 or older who are prescribed at least one medication within any of the metabolic pathways being assessed will be collected for the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Identify individual variations in metabolic pathways of 2C19, 2C9, 2D6, 3A4, 3A5, Factor II, Factor V, MTHFR and VKORC1 | 18 months
  Patients with variations in metabolic pathways of 2C19, 2C9, 2D6, 3A4, 3A5, Factor II, Factor V, MTHFR and VKORC1 that may inhibit the normal metabolism of medications that are metabolized through these pathways will be identified and care received observed for changes in healthcare plan.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Allan, Study Director — IFG Medical
Locations (1):
- Sevierville Foot and Ankle Clinic, Sevierville, Tennessee, United States

REFERENCES:
- See also: Website for site members and investigators to obtain information about opportunity. — http://bracaneco.com